CLINICAL TRIAL: NCT00954499
Title: Reducing Pain in Four- to Six-month Old Infants Undergoing Immunization Using a Multi-modal Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Janet Probst, Family Practice Nurse, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-0019
Record Dates: First submitted 2009-07-22; First posted 2009-08-07 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Pain From Immunization
Keywords: tactile stimulation; pain; immunization; infant
MeSH Terms: conditions — Pain | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (Active Comparator)
  Interventions: Behavioral: Standard care
- Tactile stimulation (Experimental)
  Interventions: Behavioral: Tactile stimulation added to Standard care

INTERVENTIONS:
Behavioral: Tactile stimulation added to Standard care — * Parent rubs the infant's skin near the injection site just before, during and after the injection.
  * Fast injection technique without aspiration.
  * Oral sucrose 2 minutes before first injection.
  * Parent holds infant close.
  Arms: Tactile stimulation
Behavioral: Standard care — * Fast injection technique without aspiration.
  * Oral sucrose 2 minutes before first injection.
  * Parent holds infant close.
  Arms: Standard care

SUMMARY:
The aim of this study is to answer the following question: In healthy infants aged four to six months undergoing routine immunization for diphtheria, tetanus, acellular pertussis, inactivated poliovirus and Haemophilus influenzae type B (DTaP-IPV-Hib) and pneumococcal conjugate vaccine (PCV) while receiving a combination of proven analgesic interventions (least painful injection technique, holding by parent, and oral sucrose solution) and non-procedural talk by the parent, does the addition of rubbing near the site of injection reduce pain as measured by the Modified Behavioral Pain Scale (MBPS) to a greater extent than no rubbing?

DETAILED DESCRIPTION:
Immunization is a significant source of pain and distress for infants. At present pain-relieving interventions are rarely employed to manage this pain.

There are many non-pharmacological methods that can be used to reduce immunization pain. These include: sugar water, fast injection without aspiration, holding infants during the procedure, and non-procedural related parental behaviours such as distraction. At present, there are no studies of tactile stimulation during noxious procedures in infants and its effectiveness, therefore, is unclear. Light rubbing of the skin near the injection site that is administered by a parent immediately before, during and immediately after immunization is an easily learned, cost neutral intervention that could offer improved pain management.

ELIGIBILITY:
Inclusion Criteria:

* healthy infants
* 4 to 6 months old
* routine immunization with DTaP-IPV-Hib and PCV

Exclusion Criteria:

* impaired neurological development
* history of seizure
* use of topical local anaesthetics at the injection site
* use of sedatives or narcotics in the preceding 24 hours
* fever or illness that would prevent administration of the vaccine
* parent is unable to use the assessment tools in the study
* parent does not speak English
* prior participation in this trial

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Pain response to immunization, as measured by the Modified Behavioral Pain Scale (MBPS). | at time of injection on day 1

SECONDARY OUTCOMES:
Pain response to immunization as measured by observer Visual Analogue Scale (VAS). | at time of injection on day 1

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, B.Sc.Phm, M.Sc., Ph.D., Principal Investigator — University of Toronto
Locations (1):
- Women's College Hospital Family Practice Health Centre, Toronto, Ontario, Canada